CLINICAL TRIAL: NCT03046901
Title: Oral Vancomycin Treatment in Recurrent Primary Sclerosing Cholangitis in Liver Transplant Recipients
Brief Title: Vancomycin Treatment in Recurrent PSC in Liver Transplant Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: 0 subjects enrolled
Sponsor: Ochsner Health System (Other)
Responsible Party: Principal Investigator, Shamita Shah, Principal Investigator, Ochsner Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro00013111
Record Dates: First submitted 2017-01-31; First posted 2017-02-08 (Estimated); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Primary Sclerosing Cholangitis; Post- Orthotopic Liver Transplantation
Keywords: Vancomycin; Primary Sclerosing cholangitis; Post-liver transplantation
MeSH Terms: conditions — Cholangitis, Sclerosing | interventions — Vancomycin

STUDY DESIGN:
Intervention Model Description: The study will be conducted as a prospective open-label pilot study of up to 20 patients who will receive oral vancomycin for 3-12 months as treatment for recurrent PSC after liver transplantation. There will be no masking or randomization.

ARMS (1):
- Vancomycin group (Experimental): It is a single arm open label study and will constitute only one group that will be taking vancomycin for recurrent PSC post liver transplantation.
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Vancomycin — Vancomycin belongs to the family of medicines called antibiotics.When taken by mouth, is used to treat Clostridium difficile-associated diarrhea (also called C diff). C diff is a type of bacteria that causes severe diarrhea. Oral Vancomycin is also used to treat enterocolitis caused by a certain bacteria (e.g., Staphylococcus aureus). Subjects enrolled in the study will take 500 mg capsule, 3 times per day for 3-12 weeks.
  Other Names: Vancocin

SUMMARY:
The purpose of the study is to investigate the safety and efficacy of oral vancomycin in patients with recurrent Primary Sclerosing Cholangitis (PSC) after liver transplantation. The primary endpoint is looking at the effect of the drug on liver function tests, an important surrogate of PSC disease activity at 12 weeks on treatment. Secondary endpoints include a decrease in liver function tests at 1 year, changes in bilirubin and adverse events. Effective treatment at the onset of PSC recurrence may lead to decreases in disease progression, recurrent liver failure, and repeat liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. History of prior orthotopic liver transplant or liver and kidney transplant.
2. Recurrent PSC confirmed by clinical labs (AST/ALT greater than 19 or ALKP greater than normal), imaging (MRCP or ERCP), and/or liver biopsy consistent with recurrent PSC.
3. No clinical evidence of liver transplant rejection and stability of post-transplant immune suppression dosing for three months prior to enrollment in the study
4. No changes to therapy for inflammatory bowel disease for at least three months prior to enrollment (for patients with history of IBD)
5. Patients on ursodiol must have been on a stable dose for two weeks prior to enrollment and dose must be stable for the remainder of the clinical trial.
6. All patients with inflammatory bowel disease must have had a colonoscopy within a year prior to enrollment
7. No antibiotics for 2 months before starting vancomycin
8. No probiotics for 1 month prior to starting vancomycin or during study period

Exclusion Criteria

1. Allergy to vancomycin
2. Pre-existing advanced malignancies
3. Pregnancy or Lactation
4. Inability to provide consent
5. Findings suggestive of liver disease of other etiology such as chronic alcoholic liver disease, chronic hepatitis B or C infection, autoimmune hepatitis, primary biliary cirrhosis, hemochromatosis, Wilson's disease, or congenital biliary disease.
6. Current biliary obstruction
7. Active infection
8. Involvement in any other investigational study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-12-07 (Actual); Primary Completion 2019-02-25 (Actual); Study Completion 2019-02-25 (Actual)

PRIMARY OUTCOMES:
Liver Function Test | 12 weeks
  Alkaline Phosphatase (ALKP) +/- Alanine Transaminase (ALT)

SECONDARY OUTCOMES:
Liver Function Test | 1 year
  Alkaline Phosphatase (ALKP) +/- Alanine Transaminase (ALT)
Liver Function Test | 1 year
  Bilirubin

CONTACTS AND LOCATIONS:
Locations (1):
- Ochsner Medical Center, New Orleans, Louisiana, United States